CLINICAL TRIAL: NCT06452745
Title: Early Diagnosis of Colorectal Cancer Based on a Non-invasive Metabolomics Profile
Acronym: EarlyCRC
Status: Recruiting | Type: Observational
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Principal Investigator, Raquel Cumeras, Principal Investigator, Institut Investigacio Sanitaria Pere Virgili
Other Study IDs: 114/2019
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer; Colorectal Adenoma; Colorectal Polyp; Healthy
Keywords: screening; urine; fobt; biomarkers; metabolomics
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy; Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine and FOBT samples collected before colonoscopy and before colon diet preparation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Colorectal Cancer: Diagnosed colorectal cancer after histopathological analysis of biopsy and polypectomy pieces taken within a colonoscopy.
  Interventions: Procedure: Colonoscopy; Other: Urine and FOBT collection
- Adenomatous high risk polyps: Diagnosed adenomatous high risk polyps after histopathological analysis of biopsy and polypectomy pieces taken within a colonoscopy. With = or > 10 adenomas or serrated polyps and/or any sessile or flat lesion of = or >20 mm (pediculated = or >20 mm are not high risk).
  Interventions: Procedure: Colonoscopy; Other: Urine and FOBT collection
- Adenomatous medium risk polyps: Diagnosed adenomatous medium risk polyps after histopathological analysis of biopsy and polypectomy pieces taken within a colonoscopy. With 5 to 9 non-advanced serrated adenomas or polyps and/or at least 1 advanced lesion (adenoma >10mm and/or hairy component and/or high-grade dysplasia or serrated polyp >10mm and/or dysplasia).
  Interventions: Procedure: Colonoscopy; Other: Urine and FOBT collection
- Adenomatous low risk polyps: Diagnosed adenomatous low risk polyps after histopathological analysis of biopsy and polypectomy pieces taken within a colonoscopy. With 1 to 4 non-advanced adenomas (<10mm, without hairy component or high-grade dysplasia) or non-advanced serrated polyps (<10mm, without dysplasia).
  Interventions: Procedure: Colonoscopy; Other: Urine and FOBT collection
- Healthy: No luminal lesions are observed during the colonoscopy.
  Interventions: Procedure: Colonoscopy; Other: Urine and FOBT collection

INTERVENTIONS:
Procedure: Colonoscopy — Colonoscopy performed as a regular practice during colorectal cancer screening.
Other: Urine and FOBT collection — After patients agreement, urine and FOBT are collected before the colonoscopy and before the diet preparation of the colon.

SUMMARY:
Colorectal cancer is the most frequent tumor in our environment if both sexes are considered together. Every year almost 800 cases are diagnosed in the districts of Tarragona. A little more than half of colorectal cancers are cured with surgery, with or without the addition of complementary treatments with chemotherapy and/or radiation therapy. Those who are not cured is because at the time of diagnosis the disease has already spread or they spread after having been treated surgically with curative intent.

The purpose of the EarlyCRC project is to determine whether metabolites (substances of low molecular weight) can be found in the urine and stool of patients with colorectal cancer or polyps that can be easily and cheaply differentiated (urine or stool analysis) between the patients affected by colorectal cancer or polyps, from healthy individuals. For the identification of these possible metabolites, the urine analysis will be performed using the usual techniques in metabolomics, which studies the existing metabolites in biological processes.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the most frequent neoplasm in our environment if both sexes are considered together. It is the second most common neoplasm in women, after breast cancer, and the second most common in men after prostate cancer. In terms of mortality, CRC is the second leading cause of cancer death in men, after lung cancer, and second in women after breast cancer. For the year 2013, 735 cases and 262 deaths from colorectal cancer were estimated in the province of Tarragona. Since 1982, incidence rates have increased annually by more than 3% in men and by almost 2% in women. It is estimated that if no early diagnosis program was carried out, in 2020 about 900 new cases of CRC would be diagnosed, and about 300 deaths would occur1.

These figures vary according to one or other geographical areas of the world. If we consider the European population as a whole, colorectal cancer is the third most common tumor for both sexes together, after breast cancer and prostate cancer. It is the third most common tumor in men, after prostate cancer and lung cancer, and the second most common in women, after breast cancer. The mortality figures in Europe place colorectal cancer in third place for both sexes together, after lung and breast cancer, so that in men it is surpassed only by lung cancer and in women by breast cancer2 .

As in the vast majority of cancers, age is the main non-modifiable risk factor for colon and rectal cancer. More than 90% of cases are diagnosed in people over 50 years old. There is an increased risk of CRC in those with hereditary diseases such as familial colonic polyposis or Lynch syndrome, although the vast majority of colorectal cancers (more than 90% of cases) do not have a hereditary component. With respect to the modifiable risk factors, one of the most important is the consumption of red and processed meat, or meat that is heavily cooked or cooked in direct contact with fire. On the other hand, fiber, fruit and vegetable consumption, as well as dairy and micronutrients such as folate and calcium, are protective against this cancer. All these dietary factors affect the risk of the appearance of the precursor lesions of cancer, colorectal adenomas. Obesity is another risk factor, and exercise and physical activity act as protectors. Thus, CRC is considered to be caused by a combination of genetic and environmental factors, which lead to the appearance of adenomatous polyps as a premalignant lesion, and which over time acquire new mutations in their genetic material until become an adenocarcinoma1,3.

The early diagnosis of cancer and, more specifically, that of colorectal cancer, aims to detect colorectal tumors in the initial stages as well as premalignant lesions, colonic polyps. As with all neoplastic diseases, the stage at the time of diagnosis is the most important prognostic factor when it comes to survival. In this way, it has been shown that a test capable of easily and minimally invasively diagnosing the initial stages of colorectal cancer can reduce mortality from this tumor by 15-20% in program participants4. The fact of being able to detect benign polyps not only reduces mortality from colorectal cancer, but also decreases its incidence, since the removal of polyps prevents their subsequent malignancy. Currently, the test used in the early diagnosis of colorectal cancer is the determination of occult blood in faeces from the age of 50, every two years. In the event that the test comes out positive, the patient is subsequently subjected to a colonoscopic study. Collection of the faecal sample by itself may have low acceptance and therefore may compromise population participation in screening. A urine test, with an easier and "cleaner" collection technique, could be an added advantage in an early diagnosis program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a positive FOBT test result from the Colorectal Cancer Early Detection Program and referred for a colonoscopy.

Exclusion Criteria:

* Patients diagnosed with another primary neoplasm in the last 5 years, with the exception of carcinoma in situ of the cervix or non-melanoma skin cancer.
* Patients with severe kidney disease stage IV (creatinine clearance < 30 ml/min).
* Patients with severe active liver disease (hepatitis, cirrhosis).
* Refusal to sign informed consent.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort subject to the study are patients participating in the population screening program for colorectal cancer with a positive fecal occult blood test (FOBT) who are called to undergo a colonoscopy.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-07-20 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2040-06-30 (Estimated)

PRIMARY OUTCOMES:
Colonoscopy results | 3 months
  Histopathological analysis of biopsy and polypectomy pieces.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital Universitari Joan XXIII, Tarragona, Tarragona

IPD SHARING:
Plan to Share IPD: No